CLINICAL TRIAL: NCT00368017
Title: Metabolic Effects of Thiazolidinediones in Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to replace Fellow conducting the study who left institution in 2007
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060042
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: pioglitazone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — 30 mg once a day for 12 weeks
  Other Names: ACTOS
  Arms: 1
Drug: placebo — 1 pill once a day for 12 weeks
  Arms: 2

SUMMARY:
The substantially increased cardiovascular morbidity and mortality rates in chronic kidney disease (CKD) patients cannot be sufficiently explained by traditional coronary risk factors. It is apparent that inflammation of the vessel wall plays an essential role in the pathophysiology of atherosclerosis, and the strong association between elevated inflammatory biomarkers and cardiovascular death further supports this mechanism. Approximately 50% of the mortality in this population of patients is attributable to cardiovascular disease. Insulin resistance is also a common problem in uremic patients. It has been shown that insulin resistance may contribute to atherosclerotic cardiovascular disease. An intriguing observation in CKD patients with advanced uremia is that the metabolic profile of these patients is characterized by persistent low-grade inflammation, a state of insulin resistance, and significantly increased prevalence of atherosclerosis. It is possible that these metabolic derangements can be the inciting factors for development and progression of uremic atherosclerosis. Peroxisome proliferator-activated receptor gamma (PPAR-gamma) is a ligand-activated nuclear transcription factor found in cells of the immune system and the vasculature, where it exerts an overall protective effect on the development of atherosclerosis, in part through modulation of inflammation. The agonists for PPAR-gamma improve not only the insulin resistance, but also have profound beneficial effects on inflammation, oxidative stress, endothelium, and lipid metabolism. In this proposal, the investigators hypothesize that short-term administration of a PPAR-gamma agonist (pioglitazone) will improve the inflammatory state, insulin resistance, and endothelial dysfunction in chronic kidney disease patients with advanced uremia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage 3 or 4 chronic kidney disease as measured by a Modification in Diet in Renal Disease Study (MDRD) estimate of between 15 ml/min and 59 ml/min.
2. Age between 18 and 75 years old.
3. Patients without hospitalization for cardiac or infection related morbidity over the previous four weeks (due to the potential confounding effects on baseline study variables).
4. Patients who are able to provide consent to participate in the study.

Exclusion Criteria:

1. Patients with prior documented diagnosis of diabetes mellitus.
2. Patients with fasting blood glucose > 110mg/dL.
3. Prisoners, patients will significant mental illness, pregnant women, and other vulnerable populations.
4. Patients with active hepatic disease and/or ALT > 2.5 times upper limit of normal.
5. Patients with history of congestive heart failure and NYHA Class III-IV symptoms at any time.
6. Patients for whom living donor renal transplantation is already scheduled or in the process of being evaluated, as these patients will be unlikely to complete study protocols before transplantation.
7. Patients with severe co-morbid conditions (eg, symptomatic hepatic cirrhosis, metastatic cancer, HIV infection with AIDS).
8. Patient with active inflammatory process (eg., SLE, rheumatoid arthritis, gout) for which they are currently receiving immune modulating medications.
9. Patients who are on corticosteroid therapy.
10. Patients who do not consent to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
A decrease in C-reactive protein (CRP) levels | 14 weeks

SECONDARY OUTCOMES:
Improved insulin resistance | 14 weeks
Improved endothelium-dependent vasodilation | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States